CLINICAL TRIAL: NCT06978179
Title: Ultrasound-Guided Quadratus Lumborum Block Versus Transversus Abdominis Plane Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients, Prospective, Comparative Randomized Study
Brief Title: Ultrasound-Guided QL Block Versus TAP Block For Post-Operative Pain In Lower Abdominal Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Aboelnaga, Resident, Anesthesiology, Surgical ICU and Pain Medicine, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-4-01MS
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US Guided QL Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients (Active Comparator): Group ( 1 ) QLB "Type III": Patients will receive QLB performedwith20ml of diluted bupivacaine 0.25% on each side.
  Interventions: Procedure: Ultrasound-Guided Quadratus Lumborum Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients
- US Guided TAP Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients (Active Comparator): Group ( 2 ) TAP: Patients will receive TAP block performed with 20ml of diluted bupivacaine 0.25% on each side.
  Interventions: Procedure: Ultrasound-Guided Transversus Abdominis Plane Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients

INTERVENTIONS:
Procedure: Ultrasound-Guided Quadratus Lumborum Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients — Group ( 1 ) QLB "Type III": Patients will receive QLB performedwith20ml of diluted bupivacaine 0.25% on each side.
  Arms: US Guided QL Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients
Procedure: Ultrasound-Guided Transversus Abdominis Plane Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients — Group ( 2 ) TAP: Patients will receive TAP block performed with 20ml of diluted bupivacaine 0.25% on each side.
  Arms: US Guided TAP Block For Post-Operative Pain In Lower Abdominal Surgeries In Adult Patients

SUMMARY:
This study aims to compare the efficacy of ultrasound-guided QL block and TAP block for postoperative pain management following lower abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 65 years old.
* American Society of Anesthesiologists (ASA) physical status I - II.
* Patients scheduled for elective lower abdominal surgery.

Exclusion Criteria:

* Patient refusal.
* Patients with BMI (body mass index) > 35 kg.m-2 , [morbid obesity].
* Patients with significant neurological, psychatric or neuromascular disease.
* Patients had local skin infection at the block injection site.
* Patients who operated under epidural and patient-controlled analgesia [PCA].
* Sensitivity to prescribed analgesia.
* Coagulopathies or those who had uncontrolled chronic medical disease [e.g. diabetes mellitus, hypertension, or cardiac diseases].

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
efficacy of ultrasound-guided QL block and TAP block for postoperative pain management following lower abdominal surgeries. | 48 hours after operation
  Visual Analog Scale (VAS) at rest and at movement

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Borglum J, Gogenur I, Bendtsen TF. Abdominal wall blocks in adults. Curr Opin Anaesthesiol. 2016 Oct;29(5):638-43. doi: 10.1097/ACO.0000000000000378. PMID 27429253
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Chen Q, Beal EW, Okunrintemi V, Cerier E, Paredes A, Sun S, Olsen G, Pawlik TM. The Association Between Patient Satisfaction and Patient-Reported Health Outcomes. J Patient Exp. 2019 Sep;6(3):201-209. doi: 10.1177/2374373518795414. Epub 2018 Aug 27. PMID 31535008